CLINICAL TRIAL: NCT01342484
Title: A Randomised, Double-blind, Placebo-controlled, Parallel Group Dose-finding Study of Linagliptin (1 and 5 mg Administered Orally Once Daily) Over 12 Weeks in Children and Adolescents, From 10 to 17 Years of Age, With Type 2 Diabetes Mellitus
Brief Title: Finding a Safe and Effective Dose of Linagliptin in Pediatric Patients With Type 2 Diabetes
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1218.56; 2009-017004-91 (EudraCT Number: EudraCT)
Record Dates: First submitted 2011-04-26; First posted 2011-04-27 (Estimated); Results first posted 2016-09-15 (Estimated); Last update posted 2016-09-15 (Estimated); Status verified 2016-07

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Linagliptin

ARMS (3):
- linagliptin low dose (Experimental): linagliptin low dose for children once daily
  Interventions: Drug: BI1356 low dose
- linagliptin high dose (Experimental): linagliptin high dose for children once daily
  Interventions: Drug: BI1356 high dose
- placebo (Placebo Comparator): matching placebo for each linagliptin dose once daily
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: placebo — comparison of different dosages of drug (low vs high) vs placebo
  Arms: placebo
Drug: BI1356 low dose — comparison of different dosages of drug (low vs high) vs placebo
  Arms: linagliptin low dose
Drug: BI1356 high dose — comparison of different dosages of drug (low vs high) vs placebo
  Arms: linagliptin high dose

SUMMARY:
The main objective of this study is to identify the dose of linagliptin in paediatric patients.

Other efficacy objectives include the comparison of the lowering effect of linagliptin low dose, high dose and placebo on the fasting plasma glucose (FPG) observed after 12 wk of treatment.

Furthermore, the study will investigate the pharmacokinetics (PK), the pharmacodynamics (PD) and the PK/PD relationship of linagliptin in the paediatric population.

ELIGIBILITY:
Inclusion criteria:

1. Paediatric patients (children and adolescents), aged 10 to 17 years with documented diagnosis of type 2 diabetes mellitus
2. Insufficient glycaemic control (i.e. an HbA1c > 6.5% and <= 10.5%) despite treatment with diet and exercise and/or metformin (>= 1000 mg per day (or the maximum tolerated dose) at a stable dose or dosing frequency for 8 weeks prior to randomisation) and/or concomitant stable basal insulin (total daily dose must be <= 0.5U/kg with less than 10% of weekly dose change for 12 weeks prior to randomisation)
3. Negative for islet cell antigen (ICA) auto-antibodies and glutamic acid decarboxylase (GAD) auto-antibodies
4. C-peptide levels (serum) >= 1.5 ng/ml (at 90 min following a Boost challenge)

Exclusion criteria:

1. History of acute metabolic decompensation, such as diabetic ketoacidosis, within 3 months
2. Current short-acting insulin or having received short-acting insulin for more than 3 days within 1 month prior to randomisation
3. Treatment with weight reduction medications (including anti-obesity treatments)

Ages: 10 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2011-04; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (25):
- United States (2):
  - 1218.56.01006 Boehringer Ingelheim Investigational Site, San Antonio, Texas
  - 1218.56.01004 Boehringer Ingelheim Investigational Site, Norfolk, Virginia
- 1218.56.11001 Boehringer Ingelheim Investigational Site, Montreal, Quebec, Canada
- France (2):
  - 1218.56.33003 Boehringer Ingelheim Investigational Site, Fort de France Cedex
  - 1218.56.33006 Boehringer Ingelheim Investigational Site, Rouen
- Guatemala (2):
  - 1218.56.50202 Boehringer Ingelheim Investigational Site, Guatemala City
  - 1218.56.50203 Boehringer Ingelheim Investigational Site, Guatemala City
- 1218.56.39005 Boehringer Ingelheim Investigational Site, Florence, Italy
- Mexico (5):
  - 1218.56.52008 Boehringer Ingelheim Investigational Site, Chihuahua City
  - 1218.56.52002 Boehringer Ingelheim Investigational Site, Guadalajara
  - 1218.56.52001 Boehringer Ingelheim Investigational Site, León
  - 1218.56.52003 Boehringer Ingelheim Investigational Site, Monterrey
  - 1218.56.52004 Boehringer Ingelheim Investigational Site, Oaxaca City
- Poland (4):
  - 1218.56.48002 Boehringer Ingelheim Investigational Site, Gdansk
  - 1218.56.48001 Boehringer Ingelheim Investigational Site, Gliwice
  - 1218.56.48004 Boehringer Ingelheim Investigational Site, Warsaw
  - 1218.56.48003 Boehringer Ingelheim Investigational Site, Wroclaw
- Russia (4):
  - 1218.56.70001 Boehringer Ingelheim Investigational Site, Moscow
  - 1218.56.70003 Boehringer Ingelheim Investigational Site, Saratov
  - 1218.56.70004 Boehringer Ingelheim Investigational Site, Ufa
  - 1218.56.70006 Boehringer Ingelheim Investigational Site, Yekaterinburg
- South Korea (4):
  - 1218.56.82005 Boehringer Ingelheim Investigational Site, Busan
  - 1218.56.82001 Boehringer Ingelheim Investigational Site, Seoul
  - 1218.56.82002 Boehringer Ingelheim Investigational Site, Seoul
  - 1218.56.82003 Boehringer Ingelheim Investigational Site, Suwon

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Randomised, double-blind, placebo-controlled parallel group dose-finding study of linagliptin over 12 weeks in children and adolescents, from 10 to 17 years of age, with type 2 diabetes mellitus. Due to serious Good clinical practice (GCP) breach, 1 patient excluded from all analyses. So protocol section has 40 subjects and participant flow has 39
Pre-assignment Details: All patients suitable after screening underwent a 2-week open-label placebo run-in period before randomisation. Patients who successfully completed this period and who still met the inclusion/exclusion criteria were randomised to the 12-week randomised period in which they received either 1 of the 2 doses of linagliptin or placebo.
Groups:
- Placebo: Matching placebo dose was administered orally once daily for 12 weeks
- Linagliptin 1 mg: Linagliptin 1 mg dose was administered orally once daily for 12 weeks
- Linagliptin 5 mg: Linagliptin 5 mg dose was administered orally once daily for 12 weeks
Period: Overall Study
Arm/Group | Placebo | Linagliptin 1 mg | Linagliptin 5 mg
Started | 15 | 10 | 14
Completed | 13 | 10 | 13
Not Completed | 2 | 0 | 1
Not completed — Other Reasons | 1 | 0 | 0
Not completed — Protocol Violation | 0 | 0 | 1
Not completed — Withdrawal by Subject | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Treated set (TS) including all patients who were treated with at least one dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Linagliptin 1 mg | Linagliptin 5 mg | Total
Number analyzed (Participants) | 15 | 10 | 14 | 39
Age, Continuous [Mean (Standard Deviation); unit: Years] | 13.7 (2.0) | 14.0 (1.8) | 14.3 (2.1) | 14.0 (1.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 4 | 9 | 21
  Male | 7 | 6 | 5 | 18

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Glycosylated Haemoglobin (HbA1c) (%) After 12 Weeks of Treatment
Description: Change from baseline in Glycosylated haemoglobin (HbA1c) [%] after 12 weeks of treatment with double-blind trial medication. Baseline was defined as the last observation before the first intake of any double-blind randomised trial medication. The number of participants analysed displays the number of participants with available data at the timepoint of interest.
Time Frame: Baseline and 12 weeks
Population: Full analysis set (FAS) including all randomised patients who were treated with at least one dose of study drug and had a baseline and at least one on-treatment HbA1c assessment. Observed Case (OC): In the OC analysis, values after the use of rescue medication were set to missing.
Measure: Least Squares Mean (Standard Error); unit: Percentage of HbA1c
Arm/Group | Placebo | Linagliptin 1 mg | Linagliptin 5 mg
Number analyzed (Participants) | 11 | 8 | 13
Percentage of HbA1c | 0.45 (0.31) | -0.03 (0.38) | -0.19 (0.30)
Statistical Analysis 1: Comparison: Placebo vs Linagliptin 1 mg; Superiority of Linagliptin 1 mg vs. placebo: change from baseline in HbA1c using a restricted maximum likelihood (REML) - based mixed model repeated measures (MMRM) approach. Model includes baseline HbA1c and age as linear covariates; treatment, gender, pharmacokinetic (PK) / pharmacodynamics (PD) subgroup, background therapy, visit and visit by treatment interaction as fixed effects and patient as a random effect. The unstructured covariance structure has been used to fit the mixed model; Test type: Superiority or Other; p = 0.3295, Mixed Models Analysis; The Kenward-Roger approximation was used to estimate denominator degrees of freedom; Mean Difference (Net) = -0.48, 95% CI 2-sided [-1.47 to 0.51], Standard Error of Mean 0.48 — Mean Difference (Net Values) is actually the adjusted mean difference calculated as Linagliptin 1 mg minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Linagliptin 5 mg; Superiority of Linagliptin 5 mg vs. placebo: change from baseline in HbA1c using a restricted maximum likelihood (REML) - based mixed model repeated measures (MMRM) approach. Model includes baseline HbA1c and age as linear covariates; treatment, gender, PK/PD subgroup, background therapy, visit and visit by treatment interaction as fixed effects and patient as a random effect. The unstructured covariance structure has been used to fit the mixed model; Test type: Superiority or Other; p = 0.1447, Mixed Models Analysis; The Kenward-Roger approximation was used to estimate denominator degrees of freedom; Mean Difference (Net) = -0.63, 95% CI 2-sided [-1.50 to 0.23], Standard Error of Mean 0.42 — Mean Difference (Net Values) is actually the adjusted mean difference calculated as Linagliptin 5 mg minus Placebo

2. Secondary Outcome: Dipeptidyl-peptidase-4 (DPP-4) Inhibition (%) at Trough at Steady State
Description: DPP-4 inhibition (%) at trough at steady state is the relative change between the measurement of DPP-4 activity taken 0.5 hours before dosing at baseline and the first available on-treatment measurement of DPP-4 activity taken 0.5 hour before dosing at week 4, 8 or 12: DPP-4 inhibition (%) = 100 - (DPP-4 activity at week X / DPP-4 activity at baseline) x 100.
Time Frame: Baseline and 4 weeks or 8 weeks or 12 weeks
Population: Full analysis set (FAS) including all randomised patients who were treated with at least one dose of study drug and had a baseline and at least one on-treatment HbA1c assessment. OR (Original Results). The analysis excludes placebo patients and 1 FAS patient from Linagliptin 1 mg group.
Measure: Median (Inter-Quartile Range); unit: Percentage of DPP-4 inhibition
Arm/Group | Placebo | Linagliptin 1 mg | Linagliptin 5 mg
Number analyzed (Participants) | 0 | 9 | 13
Percentage of DPP-4 inhibition |  | 38.4 [26.9 to 48.8] | 78.9 [67.7 to 84.0]

3. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose (FPG) After 12 Weeks of Treatment
Description: Change from baseline in FPG (mmol/L) after 12 weeks of treatment with double-blind trial medication. The number of participants analysed displays the number of participants with available data at the timepoint of interest.
Time Frame: Baseline and 12 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | Placebo | Linagliptin 1 mg | Linagliptin 5 mg
Number analyzed (Participants) | 12 | 8 | 13
mmol/L | 1.70 (0.85) | 1.39 (1.07) | -0.19 (0.83)
Statistical Analysis 1: Comparison: Placebo vs Linagliptin 1 mg; Superiority of Linagliptin 1 mg vs. placebo: change from baseline in FPG using a restricted maximum likelihood (REML) - based mixed model repeated measures (MMRM) approach. Model includes baseline HbA1c, baseline FPG and age as linear covariates; treatment, gender, PK/PD subgroup, background therapy, visit and visit by treatment interaction as fixed effects and patient as a random effect. The unstructured covariance structure has been used to fit the mixed model; Test type: Superiority or Other; p = 0.8216, Mixed Models Analysis; The Kenward-Roger approximation was used to estimate denominator degrees of freedom; Mean Difference (Net) = -0.31, 95% CI 2-sided [-3.08 to 2.46], Standard Error of Mean 1.36 — Mean Difference (Net Values) is actually the adjusted mean difference calculated as Linagliptin 1 mg minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Linagliptin 5 mg; Superiority of Linagliptin 5 mg vs. placebo: change from baseline in FPG using a restricted maximum likelihood (REML) - based mixed model repeated measures (MMRM) approach. Model includes baseline HbA1c, baseline FPG and age as linear covariates; treatment, gender, PK/PD subgroup, background therapy, visit and visit by treatment interaction as fixed effects and patient as a random effect. The unstructured covariance structure has been used to fit the mixed model; Test type: Superiority or Other; p = 0.1189, Mixed Models Analysis; The Kenward-Roger approximation was used to estimate denominator degrees of freedom; Mean Difference (Net) = -1.90, 95% CI 2-sided [-4.31 to 0.52], Standard Error of Mean 1.18 — Mean Difference (Net Values) is actually the adjusted mean difference calculated as Linagliptin 5 mg minus Placebo

ADVERSE EVENTS:
Time Frame: From the first intake of study drug until 7 days after the last drug administration, up to 13 weeks.
Arm/Group | Placebo | Linagliptin 1 mg | Linagliptin 5 mg
Serious Adverse Events (participants affected / at risk) | 1/15 | 0/10 | 0/14
Other Adverse Events (participants affected / at risk) | 7/15 | 8/10 | 6/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=15) | Linagliptin 1 mg (N=10) | Linagliptin 5 mg (N=14)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=15) | Linagliptin 1 mg (N=10) | Linagliptin 5 mg (N=14)
Hyperthyroidism (Endocrine disorders) | 1 | 0 | 0
Eye haemorrhage (Eye disorders) | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 0
Lip oedema (Gastrointestinal disorders) | 1 | 0 | 0
Toothache (Gastrointestinal disorders) | 1 | 0 | 0
Conjunctivitis bacterial (Infections and infestations) | 0 | 1 | 0
Influenza (Infections and infestations) | 1 | 0 | 0
Nasopharyngitis (Infections and infestations) | 1 | 3 | 0
Respiratory tract infection (Infections and infestations) | 1 | 0 | 0
Vulvovaginitis (Infections and infestations) | 0 | 0 | 1
Joint injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Blood creatinine increased (Investigations) | 0 | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 2 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Dizziness (Nervous system disorders) | 0 | 1 | 0
Headache (Nervous system disorders) | 1 | 0 | 4
Paraesthesia (Nervous system disorders) | 0 | 1 | 1
Menorrhagia (Reproductive system and breast disorders) | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.